CLINICAL TRIAL: NCT00366249
Title: A Multicenter, Randomized, Double-Blind, Comparison Study of the Safety and Efficacy of a Once-Daily Dose of Tigecycline Versus Ertapenem for the Treatment of Foot Infections in Subjects With Diabetes
Brief Title: Study Evaluating the Safety and Efficacy of a Once-daily Dose of Tigecycline vs Ertapenem in Diabetic Foot Infections (DFI) With a Substudy in Patients With Diabetic Foot Infections Complicated by Osteomyelitis.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Wyeth (Registry Contact: Clinical Trial Registry Specialist), Wyeth
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 3074K5-319
Record Dates: First submitted 2006-08-17; First posted 2006-08-21 (Estimated); Results first posted 2009-08-21 (Estimated); Last update posted 2010-04-28 (Estimated); Status verified 2010-04

CONDITIONS: Bacterial Infections; Diabetic Foot; Osteomyelitis
Keywords: Diabetic foot infection; Osteomyelitis; Diabetes Complications; Foot ulcer; Skin infection
MeSH Terms: conditions — Bacterial Infections; Diabetic Foot; Osteomyelitis; Diabetes Complications; Foot Ulcer; Cellulitis | interventions — Tigecycline; Ertapenem

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Active Comparator)
  Interventions: Drug: Tigecycline
- B (Active Comparator)
  Interventions: Drug: Ertapenem

INTERVENTIONS:
Drug: Tigecycline — 150 mg Tigecycline once-daily IV infusion for up to 28 days, or 42 days for the substudy wth osteomyelitis
  Arms: A
Drug: Ertapenem — Ertapenem 1g IV infusion every 24 hours +/- vancomycin depending on culture results and at the discretion of investigator (for coverage of Methicillin-resistant Staphylococcus aureus (MRSA), coagulase-negative staphylococci (CNS) or enterococci coverage).
  Arms: B

SUMMARY:
The purpose of this study was to look at the safety and effectiveness of a once-daily dose of tigecycline compared to ertapenem for the treatment of diabetic foot infections. The co-primary efficacy endpoints were not met.

ELIGIBILITY:
Main inclusion criteria:

* Men and women aged 18 or older with diabetes and a qualifying foot infection. People with evidence of a diabetic foot infection with osteomyelitis may qualify for the osteomyelitis substudy arm.

Main exclusion criteria:

* People with additional significant disease, infection with resistant pathogens, contraindication, or hypersensitivity to any test article or related antibiotic.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1061 (Actual)
Dates: Start 2007-01; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer; Trial Manager, Principal Investigator — For Belgium, trials-BEL@wyeth.com; Trial Manager, Principal Investigator — For Hungary, WPBUMED@wyeth.com; Trial Manager, Principal Investigator — For Spain, infomed@wyeth.com; Trial Manager, Principal Investigator — For Taiwan, medinfo@wyeth.com; Trial Manager, Principal Investigator — For South Africa, ZAFinfo@wyeth.com; Trial Manager, Principal Investigator — For Canada, clintrialparticipation@wyeth.com; Trial Manager, Principal Investigator — For Australia, medinfo@wyeth.com; Trial Manager, Principal Investigator — For Austria, WPVIMED@wyeth.com; Trial Manager, Principal Investigator — For Croatia, WPBUMED@wyeth.com; Trial Manager, Principal Investigator — For Latvia, WPVIMED@wyeth.com; Trial Manager, Principal Investigator — For Lithuania, WPVIMED@wyeth.com; Trial Manager, Principal Investigator — For Romania, WVPIMED@wyeth.com; Trial Manager, Principal Investigator — For Argentina, Scheima@wyeth.com; Trial Manager, Principal Investigator — For Brazil, xavierl@wyeth.com; Trial Manager, Principal Investigator — For Chile, scheima@wyeth.com; Trial Manager, Principal Investigator — For Mexico, gomezzlj@wyeth.com; Trial Manager, Principal Investigator — For Sweden, MedInfoNord@wyeth.com; Trial Manager, Principal Investigator — For Germany, medinfoDEU@wyeth.com; Trial Manager, Principal Investigator — For Denmark, medinfonord@wyeth.com; Trial Manager, Principal Investigator — For Estonia, WVPMED@wyeth.com; Trial Manager, Principal Investigator — For Finland, MedInfoNord@wyeth.com; Trial Manager, Principal Investigator — For France, infomedfrance@wyeth.com; Trial Manager, Principal Investigator — For UK/Great Britian: ukmedinfo@wyeth.com; Trial Manager, Principal Investigator — For Switzerland, med@wyeth.com; Trial Manager, Principal Investigator — For Greece, decresg@wyeth.com; Trial Manager, Principal Investigator — For Italy, descresg@wyeth.com; Trial Manager, Principal Investigator — For Poland, WPWZMED@wyeth.com; Trial Manager, Principal Investigator — For Russia, WVPIMED@wyeth.com; Trial Manager, Principal Investigator — For Slovakia, DIS-WP-BV-EUBV01-Medical@wyeth.com; Trial Manager, Principal Investigator — For Turkey, Erisc@wyeth.com; Trial Manager, Principal Investigator — For Ukraine, WVPIMED@wyeth.com; Trial Manager, Principal Investigator — For China, medinfo@wyeth.com
Locations (167):
- United States (23):
  - Los Angeles, California
  - Northridge, California
  - San Francisco, California
  - Sylmar, California
  - Torrance, California
  - Orlando, Florida
  - Pensacola, Florida
  - West Palm Beach, Florida
  - Honolulu, Hawaii
  - Chicago, Illinois
  - Evanston, Illinois
  - North Chicago, Illinois
  - Springfield, Illinois
  - Baltimore, Maryland
  - Boston, Massachusetts
  - Somers Point, New Jersey
  - Winston-Salem, North Carolina
  - Lima, Ohio
  - Toledo, Ohio
  - West Reading, Pennsylvania
  - Columbia, South Carolina
  - Dallas, Texas
  - San Antonio, Texas
- Argentina (15):
  - Buenos Aires, Buenos Aires
  - Chivilcoy, Buenos Aires
  - Ciudadela, 3 de Febrero, Buenos Aires
  - La Plata, Buenos Aires
  - Loma Hermosa, Buenos Aires
  - Mar del Plata, Buenos Aires
  - Merlo, Buenos Aires
  - Morón, Buenos Aires
  - Paraná, Entre Ríos Province
  - Tunuyán, Mendoza Province
  - Rosario, Santa Fe Province
  - San Miguel de Tucumán, Tucumán Province
  - Buenos Aires
  - Córdoba
  - Mendoza
- Melbourne, Victoria, Australia
- Vienna, Austria
- Belgium (3):
  - Bornem
  - Brussels
  - Pellenberg
- Brazil (2):
  - Rio de Janeiro
  - São Paulo
- Canada (8):
  - Vancouver, British Columbia
  - Winnipeg, Manitoba
  - Hamilton, Ontario
  - Ottawa, Ontario
  - Chicoutimi, Quebec
  - Montreal, Quebec
  - Sherbrooke, Quebec
  - Trois-Rivières, Quebec
- Chile (2):
  - Santiago
  - Valdivia
- China (4):
  - Harbin, Heilongjiang
  - Beijing
  - Guangzhou
  - Tianjin
- Bogotá, Colombia
- Croatia (2):
  - Zadar
  - Zagreb
- Odense, Denmark
- Estonia (3):
  - Kohtla-Järve, Ida-Virumaa
  - Tallinn
  - Tartu
- Finland (2):
  - Kuopio
  - Turku
- France (2):
  - Strasbourg
  - Tourcoing
- Germany (5):
  - Giessen, Hesse
  - Bochum, North Rhine-Westphalia
  - Gelsenkirchen, North Rhine-Westphalia
  - Rheine, North Rhine-Westphalia
  - Münster, Northrhien-Westphalia
- Greece (3):
  - Athens
  - Holargos, Athens
  - Rio-Patras
- Hungary (5):
  - Budapest
  - Debrecen
  - Győr
  - Kistarcsa
  - Székesfehérvár
- India (4):
  - Vadodara, Gujarat
  - Bangalore, Karnataka
  - Pune, Maharashtra
  - Jaipur, Rajasthan
- Italy (3):
  - Abano Terme (PD)
  - Pisa
  - Rome
- Latvia (2):
  - Liepāja
  - Riga
- Lithuania (5):
  - Kaunas
  - Klaipėda
  - Panevezys
  - Šiauliai
  - Vilnius
- Mexico (8):
  - Colonia El Ritiro, Guadalajara
  - Guadalajara, Jalisco
  - Mendoza, Mendoza
  - Santa Fe, Santa Fe
  - Hermosillo, Sonora
  - Durango
  - San Luis Potosí City
  - Veracruz
- Panama City, Panama
- Lima, Peru
- Poland (6):
  - Bielsko-Biala
  - Cieszyn
  - Gdansk
  - Lodz
  - Warsaw
  - Wroclaw
- Lisbon, Portugal
- Romania (4):
  - Bacau
  - Bucharest
  - Cluj-Napoca
  - Lasi
- Russia (10):
  - Chelyabinsk
  - Kemerovo
  - Moscow
  - Nizhny Novgorod
  - Novosibirsk
  - Omsk
  - Saint Petersburg
  - Smolensk
  - Yaroslavl
  - Yekaterinburg
- Slovakia (7):
  - Banska.Bysterica
  - Banská Bystrica
  - Bratislava
  - Ľubochňa
  - Martin
  - Nitra
  - Nové Zámky
- South Africa (3):
  - Port Elizabeth, Eastern Cape
  - Benoni, Gauteng
  - Pretoria, Gauteng
- South Korea (2):
  - Gyeonggi-do
  - Seoul
- Spain (5):
  - Barcelona
  - Getafe Madrid
  - Granada
  - Madrid
  - Palma de Mallorca
- Sweden (3):
  - Copenhagen
  - Huddinge
  - Uppsala
- Switzerland (2):
  - Basel
  - Geneva
- Taiwan (2):
  - Tainan
  - Taoyuan Hsien
- Turkey (Türkiye) (3):
  - Adana
  - Capa-Istanbul
  - Istanbul
- Ukraine (7):
  - Cherkassy
  - Dnipro
  - Kiev
  - Kyiv
  - Lviv
  - Vinnytsia
  - Zaporizhzhya
- United Kingdom (5):
  - Wishaw, Lanarkshire
  - Birmingham, West Midlands
  - Birmingham
  - London
  - Oxford

REFERENCES:
- [Derived] Lauf L, Ozsvar Z, Mitha I, Regoly-Merei J, Embil JM, Cooper A, Sabol MB, Castaing N, Dartois N, Yan J, Dukart G, Maroko R. Phase 3 study comparing tigecycline and ertapenem in patients with diabetic foot infections with and without osteomyelitis. Diagn Microbiol Infect Dis. 2014 Apr;78(4):469-80. doi: 10.1016/j.diagmicrobio.2013.12.007. Epub 2013 Dec 16. PMID 24439136

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited worldwide from January 2007 to February 2009.
Pre-assignment Details: Patients were screened for up to 24 hours.
Groups:
- Tigecycline: Tigecycline 150 mg IV infusion every 24 hours
Period: Overall Study
Arm/Group | Tigecycline | Ertapenem
Started | 553 | 508
Completed | 422 | 430
Not Completed | 131 | 78
Not completed — Adverse Event | 53 | 28
Not completed — Death | 0 | 1
Not completed — Physician Decision | 5 | 2
Not completed — Lost to Follow-up | 2 | 0
Not completed — Protocol Violation | 1 | 2
Not completed — Withdrawal by Subject | 18 | 4
Not completed — Lack of Efficacy | 21 | 21
Not completed — Most due to osteomylitis status | 31 | 20

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tigecycline | Ertapenem | Total
Number analyzed (Participants) | 553 | 508 | 1061
Age Continuous [Mean (Standard Deviation); unit: years] | 59.36 (12.04) | 58.75 (11.70) | 59.07 (11.88)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 199 | 165 | 364
  Male | 354 | 343 | 697

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Clinical Response of Cure Vs. Failure.
Description: Cure: Recovery so no added antibiotic therapy. Failure: Added antibiotic therapy for no response or worsening after improvement, new purulence, >120% doses, non-routine surgical treatment or death related to Diabetic Foot Infections (DFI) > 48 hrs.
Time Frame: Test of cure visit (TOC): Assessed at least 12 days post last dose
Population: Clinically evaluable population without osteomyelitis.
Measure: Number; unit: patients
Arm/Group | Tigecycline | Ertapenem
Number analyzed (Participants) | 408 | 405
patients
  Cure | 316 | 334
  Failure | 92 | 71
Statistical Analysis 1: Comparison: Tigecycline vs Ertapenem; Analysis provided for Cure; Test type: Non-Inferiority or Equivalence — Statistical analysis tested for non-inferiority. Non-inferiority margin is -10%; Mehrotra and Railker = -5.5, 95% CI [-11.0 to 0.1] — Adjusted for Perfusion, Extent, Depth/tissue loss, Infection, and Sensation (PEDIS) score

2. Secondary Outcome: Number of Patients With Clinical Response of Cure Vs. Failure Assessed at Least 25 - 27 Weeks Post Last Dose.
Description: Cure: Recovery so no added antibiotic therapy. Failure: Added antibiotic therapy for no response or worsening after improvement, new purulence, >120% doses, non-routine surgical treatment or death related to DFI > 48 hrs.
Time Frame: Test of cure visit (TOC): Assessed at least 25 - 27 weeks post last dose
Population: Clinically evaluable population with osteomyelitis.
Measure: Number; unit: patients
Arm/Group | Tigecycline | Ertapenem
Number analyzed (Participants) | 38 | 24
patients
  Cure | 12 | 13
  Failure | 26 | 11

3. Primary Outcome: Number of Patients With Clinical Response of Cure Vs. Failure/Indeterminate.
Description: Cure: Recovery so no added antibiotic therapy. Failure: Added antibiotic therapy for no response or worsening after improvement, new purulence, >120% doses, non-routine surgical treatment or death related to DFI > 48 hrs. Indeterminate: Lost to follow-up, death<48 hours or noninfection related.
Time Frame: Test of cure visit (TOC): Assessed at least 12 days post last dose
Population: Clinical modified intent to treat population without osteomyelitis.
Measure: Number; unit: patients
Arm/Group | Tigecycline | Ertapenem
Number analyzed (Participants) | 476 | 466
patients
  Cure | 340 | 363
  Failure | 117 | 86
  Indeterminate | 19 | 17
Statistical Analysis 1: Comparison: Tigecycline vs Ertapenem; Analysis provided for Cure; Test type: Non-Inferiority or Equivalence — Statistical analysis tested for non-inferiority. Non-inferiority margin is -10%; Mehrotra and Railkar = -6.7, 95% CI [-12.3 to -1.1] — Adjusted for PEDIS score

4. Secondary Outcome: Number of Patients With Clinical Response of Cure Vs. Failure/Indeterminate Assessed at Least 25 - 27 Weeks Post Last Dose.
Description: as for outcome 3
Time Frame: Test of cure visit (TOC): Assessed at least 25 - 27 weeks post last dose
Population: Clinical modified intent to treat population with osteomyelitis.
Measure: Number; unit: patients
Arm/Group | Tigecycline | Ertapenem
Number analyzed (Participants) | 53 | 33
patients
  Cure | 19 | 21
  Failure | 27 | 12
  Indeterminate | 7 | 0

5. Secondary Outcome: Number of Patients With Microbiologic Response of Eradication.
Description: Eradication defined as: no pathogen is present in the repeat culture from the original site of infection, or a clinical response of the cure precludes the availability of a specimen for culture.
Time Frame: Test of cure visit (TOC): Assessed at least 12 days post last dose
Population: Microbiologically evaluable population without osteomyelitis.
Measure: Number; unit: patients
Arm/Group | Tigecycline | Ertapenem
Number analyzed (Participants) | 316 | 317
patients | 209 | 229
Statistical Analysis 1: Comparison: Tigecycline vs Ertapenem; Test type: Non-Inferiority or Equivalence — Statistical analysis tested for non-inferiority. Non-inferiority margin is -10%; Mehrotra and Railkar = -6.3, 95% CI [-13.6 to 1.0] — Adjusted for PEDIS score

ADVERSE EVENTS:
Arm/Group | Tigecycline | Ertapenem
Serious Adverse Events (participants affected / at risk) | 79 | 62
Other Adverse Events (participants affected / at risk) | 406 | 292
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Tigecycline | Ertapenem
Abdominal pain (General disorders) | 1/553 | 0/508
Abscess (General disorders) | 5/553 | 0/508
Accidental injury (General disorders) | 0/553 | 1/508
Allergic reaction (General disorders) | 1/553 | 0/508
Asthenia (General disorders) | 0/553 | 1/508
Carcinoma (General disorders) | 0/553 | 1/508
Cellulitis (General disorders) | 1/553 | 0/508
Chest pain (General disorders) | 2/553 | 1/508
Fever (General disorders) | 4/553 | 0/508
Gangrene (General disorders) | 3/553 | 2/508
Infection (General disorders) | 9/553 | 16/508
Pain (General disorders) | 0/553 | 1/508
Sepsis (General disorders) | 1/553 | 1/508
Septic shock (General disorders) | 1/553 | 0/508
Sudden death (General disorders) | 1/553 | 0/508
Arterial thrombosis (Vascular disorders) | 1/553 | 1/508
Atrial fibrillation (Cardiac disorders) | 2/553 | 0/508
Bundle branch block (Cardiac disorders) | 0/553 | 1/508
Cardiomegaly (Cardiac disorders) | 0/553 | 1/508
Cerebral ischemia (Cardiac disorders) | 1/553 | 0/508
Cerebrovascular accident (Cardiac disorders) | 0/553 | 2/508
Congestive heart failure (Cardiac disorders) | 1/553 | 2/508
Coronary artery disorder (Cardiac disorders) | 1/553 | 0/508
Deep vein thrombosis (Vascular disorders) | 1/553 | 0/508
Heart arrest (Cardiac disorders) | 1/553 | 0/508
Heart failure (Cardiac disorders) | 0/553 | 1/508
Hemorrhage (Vascular disorders) | 0/553 | 1/508
Myocardial infarct (Cardiac disorders) | 4/553 | 0/508
Occlusion (Cardiac disorders) | 1/553 | 2/508
Peripheral gangrene (Vascular disorders) | 2/553 | 0/508
Peripheral vascular disorder (Vascular disorders) | 1/553 | 2/508
Pulmonary embolus (Vascular disorders) | 1/553 | 0/508
Shock (Cardiac disorders) | 2/553 | 0/508
Syncope (Cardiac disorders) | 1/553 | 2/508
Tachycardia (Cardiac disorders) | 1/553 | 0/508
Thrombophlebitis (Vascular disorders) | 0/553 | 1/508
Thrombosis (Vascular disorders) | 0/553 | 1/508
Vasculitis (Vascular disorders) | 1/553 | 0/508
Cholelithiasis (Gastrointestinal disorders) | 1/553 | 0/508
Cirrhosis of liver (Gastrointestinal disorders) | 1/553 | 0/508
Diarrhea (Gastrointestinal disorders) | 1/553 | 1/508
Gastritis (Gastrointestinal disorders) | 1/553 | 0/508
Gastroenteritis (Gastrointestinal disorders) | 1/553 | 0/508
Gastrointestinal hemorrhage (Gastrointestinal disorders) | 1/553 | 0/508
Ileus (Gastrointestinal disorders) | 1/553 | 0/508
Liver damage (Gastrointestinal disorders) | 1/553 | 0/508
Nausea (Gastrointestinal disorders) | 6/553 | 0/508
Stomach atony (Gastrointestinal disorders) | 1/553 | 0/508
Vomiting (Gastrointestinal disorders) | 6/553 | 0/508
Leukocytosis (Blood and lymphatic system disorders) | 1/553 | 0/508
Neutropenia (Blood and lymphatic system disorders) | 0/553 | 1/508
Acidosis (Metabolism and nutrition disorders) | 1/553 | 0/508
Alkaline phosphatase increased (Metabolism and nutrition disorders) | 0/553 | 1/508
Dehydration (Metabolism and nutrition disorders) | 1/553 | 0/508
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0/553 | 1/508
Healing abnormal (Metabolism and nutrition disorders) | 1/553 | 1/508
Hypoglycemia (Metabolism and nutrition disorders) | 3/553 | 0/508
Hypoglycemic reaction (Metabolism and nutrition disorders) | 0/553 | 1/508
Lipase increased (Metabolism and nutrition disorders) | 1/553 | 0/508
Arthrosis (Musculoskeletal and connective tissue disorders) | 1/553 | 1/508
Osteomyelitis (Musculoskeletal and connective tissue disorders) | 17/553 | 5/508
Pyogenic arthritis (Musculoskeletal and connective tissue disorders) | 1/553 | 0/508
Convulsion (Nervous system disorders) | 2/553 | 4/508
Hallucinations (Nervous system disorders) | 0/553 | 1/508
Hypesthesia (Nervous system disorders) | 0/553 | 1/508
Mental status changes (Nervous system disorders) | 1/553 | 1/508
Neuropathy (Nervous system disorders) | 0/553 | 1/508
Somnolence (Nervous system disorders) | 1/553 | 0/508
Stupor (Nervous system disorders) | 0/553 | 1/508
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0/553 | 1/508
Aspiration pneumonia (Respiratory, thoracic and mediastinal disorders) | 0/553 | 1/508
Cough increased (Respiratory, thoracic and mediastinal disorders) | 1/553 | 0/508
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2/553 | 0/508
Lung edema (Respiratory, thoracic and mediastinal disorders) | 1/553 | 0/508
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0/553 | 1/508
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 2/553 | 1/508
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1/553 | 1/508
Skin necrosis (Skin and subcutaneous tissue disorders) | 4/553 | 3/508
Skin ulcer (Skin and subcutaneous tissue disorders) | 2/553 | 2/508
Vesiculobullous rash (Skin and subcutaneous tissue disorders) | 0/553 | 1/508
Acute kidney failure (Renal and urinary disorders) | 1/553 | 0/508
Kidney function abnormal (Renal and urinary disorders) | 0/553 | 2/508
Urinary tract infection (Renal and urinary disorders) | 1/553 | 0/508
Local reaction to procedure (General disorders) | 0/553 | 1/508
Left heart failure (Cardiac disorders) | 2/553 | 0/508
Vascular disorder general (Vascular disorders) | 1/553 | 1/508
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected / at risk:
Term (organ system) | Tigecycline | Ertapenem
Abdominal pain (General disorders) | 20/553 | 11/508
Asthenia (General disorders) | 19/553 | 8/508
Respiratory system general (Respiratory, thoracic and mediastinal disorders) | 32/553 | 29/508
Fever (General disorders) | 27/553 | 19/508
Headache (General disorders) | 26/553 | 20/508
Skin and appendages general (Skin and subcutaneous tissue disorders) | 43/553 | 28/508
Pain (General disorders) | 25/553 | 17/508
Urogenital general (Renal and urinary disorders) | 24/553 | 27/508
Hypertension (Cardiac disorders) | 36/553 | 40/508
Diarrhea (Gastrointestinal disorders) | 75/553 | 51/508
Dyspepsia (Gastrointestinal disorders) | 19/553 | 6/508
Nausea (Gastrointestinal disorders) | 227/553 | 46/508
Vomiting (Gastrointestinal disorders) | 151/553 | 25/508
Anemia (Blood and lymphatic system disorders) | 14/553 | 18/508
Hypoglycemia (Metabolism and nutrition disorders) | 50/553 | 24/508
Serum glutamic oxaloacetic transaminase (SGOT) increased (Metabolism and nutrition disorders) | 20/553 | 21/508
Serum glutamic pyruvic transaminase (SGPT) increased (Metabolism and nutrition disorders) | 19/553 | 20/508
Osteomyelitis (Musculoskeletal and connective tissue disorders) | 25/553 | 12/508
Dizziness (Nervous system disorders) | 17/553 | 10/508
Insomnia (Nervous system disorders) | 18/553 | 5/508
Infection (General disorders) | 12/553 | 19/508

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PIs agreed to allow the sponsor 60 days to review and require changes to presentations or publications but only to protect confidential information and intellectual property, and for the sponsor to file a patent application, as applicable. The PIs also agreed for data to be presented first as a joint, multi-center publication.